CLINICAL TRIAL: NCT01068353
Title: A Phase 2, Double-blind, Placebo-controlled Study of the Safety and Tolerability of Etanercept in Patients With Alzheimer's Disease
Brief Title: Safety and Tolerability of Etanercept in Alzheimer's Disease
Acronym: STEADI-09
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southampton (Other)
Collaborators: Hampshire Hospitals NHS Foundation Trust (Other); Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STEADI-09; 2009-013400-31 (EudraCT Number)
Record Dates: First submitted 2010-02-10; First posted 2010-02-12 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; Dementia; TNF-alpha; Etanercept
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Etanercept (Experimental)
  Interventions: Biological: Etanercept

INTERVENTIONS:
Biological: Etanercept — 50 mg given as a once weekly subcutaneous injection
  Other Names: Enbrel
  Arms: Etanercept
Other: Placebo — Placebo injection given once weekly
  Arms: Placebo

SUMMARY:
The primary aim of the study is to determine the safety and tolerability of etanercept in subjects with Alzheimer's Disease. The effects of etanercept on cognitive, behavioural, functional and immunological outcomes will be examined as secondary aims.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged > 54 years
* Have a minimum of 7 years of education
* Be able to hear, read, write and perform study neuropsychological tests in English
* Have adequate visual and auditory acuity to allow neuropsychological testing based on the research clinician's judgement
* Fulfil Diagnostic & Statistical Manual (DSM-IV-TR)criteria for diagnosis of dementia of the Alzheimer type
* Have a diagnosis of probable Alzheimer's Disease (National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria)
* Mini Mental State Examination (MMSE) score < 27 and > 10 points.
* To be currently taking and have been taking a cholinesterase inhibitor for a minimum period of 3 months prior to the day of inclusion into the study or to have been not been taking a cholinesterase inhibitor for a minimum period of 3 months prior to the day of inclusion into the study
* Have an informant who spends at least 24 hours per week with the patient and may be a close friend or a neighbour, not necessarily a close relative, spouse, son or daughter. He/she should be the same throughout the study and should be present at all visits. If it becomes necessary, a change of informant can be made but this must be clearly documented.

Exclusion Criteria:

* Inability or refusal to provide informed consent from patient or caregiver
* Absence of informant
* Unlikely to cooperate in the study, not able to attend scheduled examinations and visits, or not able to follow study instructions
* Participation in another study with administration of any investigational drug in the previous 3 months or already enrolled in another study
* Parkinson's Disease, Dementia with Lewy Bodies or clinically significant Parkinsonian symptoms
* Vascular disorder (modified Hachinski Ischaemic Scale score > 4)
* Recent Transient Ischaemic Attack (TIA) - within the last 3 months
* Signs of major cerebrovascular disease on MRI or CT scan, if performed prior to entry into study (i.e. presence of infarction in greater than 25% of white matter, more than 1 lacune within basal ganglia, more than 2 lacunes in white matter)
* Any other previous or ongoing chronic or recurrent disease of the central nervous system, including demyelinating disease or psychiatric diseases, that may have an impact on cognitive performance, left to the research clinician's judgement
* Any of the following laboratory abnormalities at the screening visit:

  i) Clinically significant Vitamin B12 levels less than the lower limit of normal ii) Clinically significant folate levels less than the lower limit of normal iii) Clinically significant thyroid-stimulating hormone (TSH) levels greater than the upper limit of normal and a clinically significant free thyroxine (FT4) level lower than the lower limit of normal
* Patients with previous or present history of severe or unstable medical conditions (e.g. hypertension, diabetes left to the research clinician's judgement)
* Current alcohol >35 units per week for men, or >28 units per week for women, or drug abuse at the discretion of the research clinician
* Surgical intervention planned during the study period.
* Treatment with immunosuppressive drugs and/or oral prednisone greater than 10mg/day within the past 90 days
* Treatment with Memantine within the past 3 months
* Vaccination or immunization with any live vaccine (eg: polio, rubella, yellow fever) or the pneumococcal vaccine within the past 30 days.
* Pregnancy or breast feeding.
* Severe hepatic, renal or cardiac disease.
* Previous use of a Tumour Necrosis Factor-alpha (TNFα) agent.
* Known skin photosensitivity.
* Infection in past 4 weeks or active infection.
* Heart failure: New York Heart Association (NYHA) Grade 3-4.
* History of blood disorders or current WCC ≤ 3.5 x 109/l; platelet count ≤ 100x109/l ; Hb ≤ 10g/dl.
* Active or latent tuberculosis
* Rheumatoid arthritis; psoriasis; psoriatic arthritis or ankylosing spondylitis
* Septic arthritis in past 12 months
* Sepsis of prosthesis in past 12 months
* Chronic leg ulcers
* Indwelling urinary catheter
* Pulmonary fibrosis
* History of neoplasms / malignancies in past 5 years
* Pre-malignant conditions including Barrett's oesophagus; cervical dysplasia; large bowel polyps
* Any relevant acute or chronic abnormality detected during the physical and neurological examinations. Electrocardiogram (ECG) or laboratory tests likely to interfere with the study evaluations in the research clinician's judgement
* Previous exposure to amyloid vaccines, monoclonal antibodies or intravenous immunoglobulins meant to treat Alzheimer's disease

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events and serious adverse events (the study is a Phase II safety trial) | 6 months

SECONDARY OUTCOMES:
Difference in change in Alzheimer's Disease Assessment Scale - Cognitive Section (ADAS-cog) total score between treated and placebo groups from baseline to end point at 6 months | 6 months
Difference in change in Neuropsychiatric Inventory (NPI) total score between treated and placebo groups from baseline to end point at 6 months | 6 months
Difference in change in Clinician's Global Impression of Change (CGIC) and Carer's Impression of Change (Carer-IC) total score between treated and placebo groups from baseline to end point at 6 months | 6 months
Difference in change in Mini-Mental State Examination (MMSE) total score between treated and placebo groups from baseline to end point at 6 months | 6 months
Difference in change in Sickness Behaviour Scale between treated and placebo groups from baseline to end point at 6 months | 6 months
To establish whether a pro-inflammatory baseline cytokine profile predicts better response to treatment with etanercept | 6 months
To examine the effects of etanercept on inflammatory markers in the cerebrospinal fluid (CSF) of patients with Alzheimer's disease, and the relationship of these factors with clinical outcome | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Memory Assessment and Research Centre, Moorgreen Hospital, Southampton, Hampshire, United Kingdom

REFERENCES:
- [Derived] Butchart J, Brook L, Hopkins V, Teeling J, Puntener U, Culliford D, Sharples R, Sharif S, McFarlane B, Raybould R, Thomas R, Passmore P, Perry VH, Holmes C. Etanercept in Alzheimer disease: A randomized, placebo-controlled, double-blind, phase 2 trial. Neurology. 2015 May 26;84(21):2161-8. doi: 10.1212/WNL.0000000000001617. Epub 2015 May 1. PMID 25934853